CLINICAL TRIAL: NCT07236502
Title: Moving Forward With Myeloma: A Lifestyle Intervention for Individuals With Multiple Myeloma
Brief Title: Moving Foward With Myeloma (MFM)
Acronym: MFM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Loyola University Chicago (Other)
Responsible Party: Principal Investigator, Melinda Stolley, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00040708; 1R01CA300310 (NIH)
Record Dates: First submitted 2025-11-06; First posted 2025-11-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma (MM)
Keywords: Lifestyle Intervention
MeSH Terms: conditions — Multiple Myeloma | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Waitlist Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): 16-session intervention that facilitates changes in nutrition and physical activity behaviors to promote improvements in physical function, Patient Reported Outcomes, body composition and general health. The intervention targets plant-based eating, increasing physical activity and strength training.
  Interventions: Behavioral: Immediate intervention
- Waitlist control (Active Comparator): Participants will be asked to maintain their behavior over the 16 week waitlist period and will receive weekly text message relating positive messages unrelated to lifestyle.
  Interventions: Behavioral: Immediate intervention; Other: Waitlist

INTERVENTIONS:
Behavioral: Immediate intervention — 16-session intervention that facilitates changes in nutrition and physical activity behaviors to promote improvements in physical function, Patient Reported Outcomes, body composition and general health
Other: Waitlist — Participants will be asked to maintain their behavior over the 16 week waitlist period and will receive weekly text message relating positive messages unrelated to lifestyle
  Arms: Waitlist control

SUMMARY:
The purpose of this project is to evaluate the impact of a 16-week lifestyle program that promotes changes in eating and exercise patterns. The main questions the study will answer are:

Do improvements in eating and exercise patterns lead to improved physical function, quality of life and blood biomarkers of biologial aging among individuals with multiple myeloma? Participants will complete study activities 3-4 times during the study.

1. In-person assessment to measure physical function, height/weight, body composition, and includes a blood draw
2. Surveys completed online or on paper at home

DETAILED DESCRIPTION:
The study uses a randomized, waitlist control design. Following baseline data collection, participants will be randomized to either the immediate lifestyle intervention group or the waitlist control group. Those who are randomized to the waitlist control group will receive the intervention after the 16-week data collection time point.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years)
2. Diagnosed with MM at least one year prior to study enrollment
3. Has access to a cell phone
4. Be deemed "clinically stable" by their physician guided by the following:

   1. no near-term changes in planned myeloma-directed therapy anticipated. (e.g., patient who is 3 months from autologous stem cell transplant just starting on maintenance lenalidomide is eligible since maintenance is planned therapy following transplant)
   2. no new significant myeloma symptoms (e.g., fractures) meriting changes in anti-neoplastic therapies; AND
   3. stable performance status (ECOG 0-2)
5. No reports of severe pain > Grade 3 [defined by the NCI CTCAE as tumor, neurologic, bone, or other pain interfering with self-care ADLs (bathing, dressing, toileting, continence, feeding)].
6. Able to participate in moderate PA and strength training per clinician approval and confirmed by participant
7. Able to understand and willing to sign a written informed consent document
8. English proficient for reading and writing

Exclusion Criteria:

1. Individuals with <6 months of life anticipated, coexistent amyloidosis, and/or receiving appetite stimulants will not be approached
2. Fully adherent to the ACS nutrition and physical activity guidelines
3. Currently pregnant or lactating, or anticipating pregnancy
4. On another interventional clinical trial that precludes co-enrollment
5. Psychiatric or other clinical conditions that preclude study compliance
6. Other important medical or safety considerations at the discretion of the investigator(s) and/or approving clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-12-15 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Examine the efficacy of the intervention in producing post-intervention changes in performance-based physical function | Baseline, Week 16, Week 32, Week 48
  Changes in performance-based physical function between the interventional and control groups will be measured using the Short Physical Performance Battery (SPPB), which comprises a 4-meter walk test to assess gait speed, sit-to-stand test to assess lower body strength, and standing balance tests to assess balance. Scoring for the SPPB ranges from 0 to 12; higher scores indicate higher function.

SECONDARY OUTCOMES:
Examine the efficacy of the intervention in producing post-intervention changes in patient-reported outcomes. | Baseline, Week 16, Week 32, Week 48
  Changes in patient-reported outcomes between the interventional and control groups will be measured using: the Patient Reported Outcomes Measurement Information System (PROMIS) physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, pain intensity, satisfaction with social roles and activities, instrumental support, informational support, emotional support, companionship, cognitive function and social isolation. The PROMIS measures for this study will be used in a CAT Computer adaptive format.
• Godin Leisure Physical Activity: | Baseline, Week 16, Week 32, Week 48
  A tool querying about light, moderate, strenuous activities over 7-days and one item asking about strength training
• ASA 24-hour Dietary Recall (DR). | Baseline, Week 16, Week 32, Week 48
  Supported by the National Cancer Institute's ASA24 and with administrative assistance, a minimum of 2 unannounced 24DR will be completed pre/post-intervention using the 5-pass dietary recall methodology.
• Self-Efficacy for Eating and Exercise Behaviors: | Baseline, Week 16, Week 32, Week 48
  A validated tool consisting of 12 items to assess exercise self-efficacy and 20 items to assess healthy eating and exercise self-efficacy
Fruit and Vegetable Intake - objective measure | Baseline, Week 16, Week 32, Week 48
  • Veggie meter- Participants will be asked to complete reflective spectroscopy using the Veggie Meter; a device that non-invasively measures the level of carotenoid pigments in the skin.
Outcome Expectancy. | Baseline, Week 16, Week 32, Week 48
  • Measures positive and negative outcome expectations ("I would sleep more soundly if I exercised regularly"; "Regular exercise would increase my pain.") Higher scores indicate greater positive or negative outcome expectations.
Resilience | Baseline, Week 16, Week 32, Week 48
  • The Brief Resilience Scale (BRS) is a psychological measure designed to quantify a person's ability to 'bounce back' or recover from stressful events or trauma
Body composition | Baseline, Week 16, Week 32, Week 48
  • DEXA imaging is a 10-minute, noninvasive technique that provides precise whole-body measures of fat (total and visceral) and lean mass. Certified DXA technologists will perform and analyze whole body measures using the same machine for each participant at each time point)
Objective Physical Activity. (ActivPal): | Baseline, Week 16, Week 32, Week 48
  • Participants wear this device on the right thigh, held on by a Tegaderm patch to measure PA and sedentary time. Data are downloaded using ActiLife software and will be analyzed using recommended thresholds for moderate and vigorous PA.
Lipids and Glucose | Baseline, Week 16, Week 32, Week 48
  Utilizing clinical resources at MCW or LUC phlebotomy will be performed by trained personnel to conduct fasting blood draws and blood processing according to standard procedures. Whole blood will be collected, allowed to clot for 20 mins, and centrifuged at 2,500 rpm for 20 mins. o Lipids (HDL, LDL, Total Cholesterol, Triglycerides) and glucose measures will be procured using the Choletech LDX (Abbott, Inc.)

OTHER OUTCOMES:
Inflammation | Baseline, Week 16, Week 32, Week 48
  Examine the associations between lifestyle behaviors and serum biomarkers for inflammation. Markers of inflammation including CRP, IL-6; TNF-alpha will be analyzed (blind to randomization) in batch at the end of data collection using commercially available ELISA kits. Each sample will be assayed in duplicate and repeated if variability exceeds 15%.
Biological Aging | Baseline, Week 16, Week 32
  o Biological Aging/Cellular Senescence. Additional blood samples will be collected in PAXgene RNA (2.5 mL) tubes and stored (-80° C). Cellular senescence will be assessed via transcript abundance of the p16INK4a- and p21-encoding genes (CDKN2A and CDKN1A, respectively).23-25 A priori-defined sets of genes known to be up-regulated during the DNA damage response (DDR; 30 genes; e.g., CHEK1, SIRT1, TP53, TERF2), and the senescence-associated secretory phenotype (SASP; 61 genes; e.g., IL1A, IL13, CXCL8, CSF2, VEGF) will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Stolley, PhD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Loyola University Chicago, Maywood, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified data on participant characteristics and outcomes will be shared.
Supporting Information: Study Protocol
Time Frame: Once the study is completed, de-identified data collected during the study will be made available.
Access Criteria: Once the study is completed, de-identified data collected during the study will be deposited in the Harvard Dataverse. Raw RNA-seq, alignment, and transcript data will be made available to the research community free of charge through GEO. Since the purpose of this data sharing is to answer questions in the future, your